CLINICAL TRIAL: NCT04610151
Title: The Effects of Guided Imagery on Postoperative Pain Management: A Randomized Controlled Trial
Brief Title: The Effects of Guided Imagery on Postoperative Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Leyla ZENGİN AYDIN, Assistant Professor, Dicle University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: LZA2018/5
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Healthy; Nursing Caries
Keywords: Patient; Postoperative; Pain; Visual Analogue Scale; Guided Imagery
MeSH Terms: conditions — Pain | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Intervention Model Description: The study was conducted with patients undergoing lower extremity operations between April 2018 and May 2019 at the Necip Fazıl City Hospital (Kahramanmaraş, Turkey) as a pretest-posttest study with a quasi-experimental design and a control group.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Imagery (Experimental): Guided Imagery Intervention:The pretest data of the patients with a pain score of 4 or higher according to VAS were collected. Afterwards, the experiment group patients were applied guided imagery.
  Interventions: Other: guided imagery
- No-Reflexology Application , control group. (No Intervention): No intervention was applied on the control group patients.

INTERVENTIONS:
Other: guided imagery — Guided Imagery CD: A guided imagery CD was prepared by a web designer with the recommendations of the researcher to include relaxing, soft and slow-paced, mixed nature sounds and photographs towards reducing pain in lower extremity surgical operation patients. The directives used for guidance, the audio recordings created as a result of literature review and the video lasted for 13 minutes (
  Arms: Guided Imagery

SUMMARY:
This study was conducted to determine the effects of guided imagery on postoperative pain management.

DETAILED DESCRIPTION:
The sample of the study consisted of 60 patients (30 in the experiment and 30 in the control groups) undergoing lower extremity operations at the orthopedics clinics of the Kahramanmaras Necip Fazil City Hospital. The study was conducted between April and September 2018.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at and over the age of 18
* Patients who were able to speak Turkish
* Patients who received spinal anesthesia

Exclusion Criteria:

* Patients who had not previously used guided imagery
* Patients any disease that could cause pain outside the surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
A mean total score on the Visual Analogue Scale (VAS) | first week
  A mean total score on the VAS of four and above indicates postoperative pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Leyla ZENGİN AYDIN, Diyarbakır, Sur, Turkey (Türkiye)